CLINICAL TRIAL: NCT06104397
Title: Implementation of Exercise Strategies in Parkinson's Disease: Clinical Outcomes
Brief Title: Exercise Strategies in Parkinson's Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: University of Chicago (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Northwestern Medicine (Other)
Responsible Party: Principal Investigator, Miriam Rafferty, Director of Implementation Science, Shirley Ryan AbilityLab
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STU00219116; 1R01HD110668-01 (NIH)
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
Keywords: Exercise; Physical Activity; Physical Therapy; Activity Monitoring
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: There are 3 treatment groups: 1) standard care, 2) written exercise guidance by neurologists, and 3) physical therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard Care (No Intervention): Standard care patient's with Parkinson's Disease are receiving at each site.
- Written exercise guidance by neurologist (Active Comparator): Neurologists will provide written exercise education and guidance to their patients with Parkinson's Disease.
  Interventions: Other: Written exercise guidance by neurologist
- Physical therapy (Experimental): A consultative model of physical therapy will be implemented at each site for patient's with Parkinson's Disease.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Written exercise guidance by neurologist — Neurologists will provide written exercise education and guidance to their patients with Parkinson's Disease during neurologist visits and/or in after visit summary in the patient's EMR patient portal. The research team will facilitate the development of the written exercise guidance with input and feedback from each site's neurology, clinical, and administrative teams.
  Arms: Written exercise guidance by neurologist
Other: Physical therapy — A consultative model of physical therapy - a lower dose of physical therapy focused on physical activity and exercise promotion and coaching - will be implemented into each site. In the consultative model of physical therapy, visits are scheduled around needs of the patient, however will involve 1-4 additional visits within 3 months of evaluation and is based on personal factors that influence their exercise prognosis such as self-efficacy, readiness to change, fitness level, age, health literacy, comorbidities, and Parkinson's Disease-related motor and non-motor impairments.
  Arms: Physical therapy

SUMMARY:
The goal of this clinical trial is to learn about exercise and physical activity people with Parkinson's Disease. The main questions it aims to answer are: 1) learn about the physical activity and exercise behaviors of people with Parkinson's Disease over the course of a year and 2) compare 3 exercise guidance strategies aimed to impact exercise behavior: standard care, written exercise guidance from neurologist and/or physical therapy.

During the course of the study:

1. Participants will use activity trackers and a mobile phone application to monitor their exercise participation.
2. At the same time, the research team will be working with the participant's medical teams at Northwestern Medicine and University of Chicago Medical Center to improve the way that they deliver exercise guidance using verbal instructions and encouragement, written exercise guidance, and/or physical therapy.

DETAILED DESCRIPTION:
The purpose of this study is to gain a better understanding of how people with Parkinson's disease (PD) manage their physical activity and exercise participation with different levels of support from their communities and clinicians. We will evaluate exercise and physical activity every 3 months in a cohort of people with PD from two medical centers in the Chicagoland area: Northwestern Medicine and University of Chicago Medical Center.

During this study, we will evaluate differences in 12-month physical activity trajectories between groups enrolled during each of three conditions: (1A) standard care (condition 1, year 1), (1B) written exercise guidance (condition 2, year 2), and (1C) Consultative PT (condition 3, year 3). People with PD will be enrolled each year into an activity and exercise tracking study. Participants will be tracked using a remote therapeutic monitoring platform (Datos) and commercial grade activity trackers. Research-grade actigraphy and patient reported outcome measures will be monitored every 3 months for the first year.

All participants will be enrolled in an exercise and physical activity tracking study where they can use a remote therapeutic monitoring platform (Datos Health) to share their exercise and physical activity data with their medical and rehabilitation teams at NM and UCMC. The platform allows for synchronization of patients' activity data from their fitness tracker or smartwatch to the secure cloud-based platform. The platform can summarize steps per day, activity intensity, minutes of moderate-vigorous physical activity per day based on target heart rate zones (including an ability for physical therapists to customize the target heart rate zone).

At the 2 sites of care (Northwestern Medicine and University of Chicago), participants will be recruited based on contacting consecutive patients who meet the inclusion criteria based on scheduling and EMR screening prior to their visit with their neurologists. Contacting consecutive patients will ensure greater potential equity of enrolling participants rather than only patients engaged in support groups and exercise classes. However, after 3 months of recruitment, we will conduct a preliminary analysis of the numbers, recruitment rates, and characteristics (age, sex, race, ethnicity, disease duration, education) of the enrolling participants compared to the demographics of each clinic as a whole. We will then determine if we should use targeted recruitment strategies to increase reach to specific groups or recruitment rates by doing one or more of the following: (1) sending measures through MyChart to potentially eligible patients targeting or oversampling for higher socioeconomic, race, or ethnicity diversity or (2) reaching out to local community exercise classes or support groups using emails to community advocates and flyers to increase sample size more rapidly.

Consecutive patients meeting the eligibility criteria will be approached by a site study team member. The first contact may occur before or during a medical (physician, physician assistant, nurse practitioner) visit. The electronic health record system will be used to screen participants for eligibility in the few weeks before their visit through an institutional review board-approved electronic data warehouse data waiver. Attempts will be made to contact potential participants before their appointments, with a research coordinator attempting contact at their visit if there is no response to early contacts. If time is limited during the patient's session, we will use patient portal communication and/or phone calls after their visits depending on the preferences of each site (which will be determined during the pre-implementation barrier assessment).

Screening for eligibility will occur via a combination of data available in the EMR for existing patients and a quick screening questionnaire that can be done in person or over the phone. After identifying that the participant is interested and satisfies the inclusion criteria for the study, they will be sent an e-consent. Once consent is obtained, they will work with the study team to set a time for the baseline assessment period which will include ensuring the participant has their own -wrist-worn activity tracker and is able to get commercial grade activity tracker from the research team. At baseline and every 3-months throughout the 12-month (baseline, 3-months, 6-months, 9-months, 12-months) study, participants will complete online survey assessments including demographic questionnaires, habits and perceptions of physical activity and exercise, and healthcare and exercise resource utilization. Participants will, also, wear a research-grade physical activity monitor on a belt clip around their waist for 7-consecutive days at baseline, 3-, 6-, 9-, 12-months. In addition to research-grade physical activity monitoring, participants will be asked to asked to a personal commercially available activity tracker daily which will be synced to the Datos Health app.

ELIGIBILITY:
Inclusion Criteria:

* Have a neurologist confirmed diagnosis of Parkinson's Disease
* Hoehn&Yahr Stage 1-3
* Age 18-89 years old
* Ambulatory
* Written and verbal basic English proficiency adequate for survey completion
* Have a smart phone
* Willing to sync activity tracker with Datos health app at least every 3 days
* Willing to accept Datos' Terms and Conditions

Exclusion Criteria:

* Diagnosis of dementia or mild cognitive impairment in medical record
* Uses a rollator or rolling walker for mobility
* Other comorbidities significantly limiting ability to participate in exercise >12 weeks

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Accelerometer Measures | Average 1-week MVPA measured every 3-months throughout 12-month study period
  Minutes per day of moderate to vigorous physical activity (MVPA)

SECONDARY OUTCOMES:
Steps per Day | Average 1-week step counts measured every 3-months throughout 12-month study period
  Steps per day

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Rafferty, PT, DPT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (3):
- United States (3):
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Northwestern Medicine, Lake Forest, Illinois

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the "NICHD Plans for Sharing Human and Non-Human Data and/or Biospecimens" policy, resulting data will be shared in the Data and Specimen Hub (DASH) in de-identified format. Our research results will also be made available to the public via summaries on the Shirley Ryan AbilityLab (SRAlab) website and Northwestern University's DigitalHub, a repository for scholarly output through Northwestern University developed by Galter Health Sciences Library (Northwestern).
Supporting Information: SAP
Time Frame: Data will become available following completion and analysis of research study data. Data will be stored in our laboratory data repository system and thus will be available indefinitely.
Access Criteria: Data summaries will be publicly available on the Shirley Ryan AbilityLab website and Northwestern University DigitalHub. De-identified data will, also, be shared in the Data and Specimen Hub (DASH) through the NICHD.

REFERENCES:
- [Background] Osborne JA, Botkin R, Colon-Semenza C, DeAngelis TR, Gallardo OG, Kosakowski H, Martello J, Pradhan S, Rafferty M, Readinger JL, Whitt AL, Ellis TD. Physical Therapist Management of Parkinson Disease: A Clinical Practice Guideline From the American Physical Therapy Association. Phys Ther. 2022 Apr 1;102(4):pzab302. doi: 10.1093/ptj/pzab302. PMID 34963139
- [Background] Rafferty MR, MacDonald J, Byskosh A, Sloan L, Toledo S, Marciniak C, Simuni T. Using Implementation Frameworks to Provide Proactive Physical Therapy for People With Parkinson Disease: Case Report. Phys Ther. 2019 Dec 16;99(12):1644-1655. doi: 10.1093/ptj/pzz129. PMID 31508801
- [Background] Cavanaugh JT, Ellis TD, Earhart GM, Ford MP, Foreman KB, Dibble LE. Capturing ambulatory activity decline in Parkinson's disease. J Neurol Phys Ther. 2012 Jun;36(2):51-7. doi: 10.1097/NPT.0b013e318254ba7a. PMID 22592060